CLINICAL TRIAL: NCT01374412
Title: Examination of Bone Defects and Microcirculation Using Volume Computed Tomography and Dynamic Contrast-enhanced Magnetic Resonance Imaging
Brief Title: Investigation of Bone Defects and Microcirculation With Computed Tomography and Magnetic Resonance Imaging
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: German Cancer Research Center (Other)
Collaborators: Heidelberg University (Other)
Responsible Party: Sponsor
Other Study IDs: Transregio79B8
Record Dates: First submitted 2010-04-14; First posted 2011-06-16 (Estimated); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Osteoporosis; Multiple Myeloma; Vertebral Fracture
MeSH Terms: conditions — Osteoporosis; Multiple Myeloma; Spinal Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- osteoporosis: patients with benign osteoporosis

SUMMARY:
Subject of the proposed study is the non-invasive in vivo imaging of bone, bone marrow and localized microcirculation in test animals with osteoporosis, fractures and after placement of bone substitute material with volume computed tomography (VCT) (animals only) and functional magnetic resonance imaging (MRI).

In vivo imaging by means of functional MRI and VCT is carried out in osteoporotic rats, both after the induction of fracture as well as after the placement of bone substitute material.

Furthermore, patients with asymptomatic MM are investigated with functional MR-Imaging (Dynamic Contrast Enhancement- MRI and Intravoxel incoherent motion (IVIM)-imaging) longitudinally to predict the occurrence of osteolysis and the time to progression regarding SLIM-CRAB-Criteria (Rajkumar et al., Lancet Oncology, 2014).

Hypothesis:

1. Affection of microcirculation at the junction of bone and bone substitute material can be displayed by VCT and functional MRI
2. Functional MRI has prognostic value regarding occurrence of osteolysis and progression to MM regarding SLIM-CRAB-Criteria

DETAILED DESCRIPTION:
In an experimental study, rat models were used for imaging studies employing MRI (morphological, DCE- and DWI) and VCT. Mice were not used for imaging purposes due to the small size. Rats were shown to be of optimal size for small imaging studies.

144 patients with (suspected) asymptomatic MM were recruited for dynamic contrast-enhanced MRI (DCE-MRI) and diffusion weighted imaging (DWI) of the vertebral column as well as whole-body MRI using T1tse and STIR images every 6 months until progression and/ or occurrence of first osteolysis.

While during planning and initiation of this prospective trial MM was defined by CRAB-criteria only, in 2014 the SLIM-CRAB-criteria were proposed by the International Myeloma Working Group (Rajkumar et al., Lancet Oncology, 2014) with the goal to treat patients before development of osteolysis or other CRAB-criteria. These criteria were consequently introduced in clinical practice at our institution during the observation period of this study, which affects both inclusion and progression criteria of this study. In order to obtain a conclusive cohort with homogenous inclusion and progression criteria, SLIM-CRAB-criteria where retrospectively applied to restage all patients regarding inclusion and progression to MM defined by SLIM-CRAB-criteria.

ELIGIBILITY:
Inclusion Criteria:

* benign osteoporosis

Exclusion Criteria:

* contra-indications for MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with benign osteoporosis
Sampling Method: Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2010-07; Primary Completion 2024-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Changes of microcirculation at the interface between bone and implanted xenomaterial in animal models. | VCT and MRI 2-6 weeks after xenomaterial implantation
  Characteristics of the microcirculation within and in the close proximity of the bone defect in early stages and during the healing process after the placement of bone substitute materials in animal models. Correlation of functional imaging parameters derived from DCE-MRI, DWI and VCT assessed in the bone defect area with the later stage healing processes in the affected bone.
Progression to multiple myeloma defined by SLIM-CRAB-Criteria (Rajkumar, Lancet Oncology, 2014) | At inclusion in the study and in repetitive follow up every 6 months until progression requiring therapy, until contraindications for MRI are present, until patient wishes to leave the study or until death (assessed up to 20 years)
  In the study part applying functional imaging in asymptomatic myeloma patients, progression to Multiple Myeloma defined by SLIM-CRAB-Criteria is the primary outcome measure

SECONDARY OUTCOMES:
Occurrence of osteolysis | At inclusion in the study and in repetitive follow up every 6 months until progression requiring therapy, until contraindications for MRI are present, until patient wishes to leave the study or until death (assessed up to 20 years)
  In the study part applying functional imaging in asymptomatic myeloma patients, occurrence of osteolysis in x-ray / CT imaging is the secondary outcome measure.

CONTACTS AND LOCATIONS:
Overall Officials: Reinhard Schnettler, MD, Study Chair — Gießen University, Heidelberg
Locations (1):
- German Cancer Research Center, Heidelberg, Germany

REFERENCES:
- [Background] Rajkumar SV, Dimopoulos MA, Palumbo A, Blade J, Merlini G, Mateos MV, Kumar S, Hillengass J, Kastritis E, Richardson P, Landgren O, Paiva B, Dispenzieri A, Weiss B, LeLeu X, Zweegman S, Lonial S, Rosinol L, Zamagni E, Jagannath S, Sezer O, Kristinsson SY, Caers J, Usmani SZ, Lahuerta JJ, Johnsen HE, Beksac M, Cavo M, Goldschmidt H, Terpos E, Kyle RA, Anderson KC, Durie BG, Miguel JF. International Myeloma Working Group updated criteria for the diagnosis of multiple myeloma. Lancet Oncol. 2014 Nov;15(12):e538-48. doi: 10.1016/S1470-2045(14)70442-5. Epub 2014 Oct 26. PMID 25439696
- [Derived] Wennmann M, Klein A, Bauer F, Chmelik J, Grozinger M, Uhlenbrock C, Lochner J, Nonnenmacher T, Rotkopf LT, Sauer S, Hielscher T, Gotz M, Floca RO, Neher P, Bonekamp D, Hillengass J, Kleesiek J, Weinhold N, Weber TF, Goldschmidt H, Delorme S, Maier-Hein K, Schlemmer HP. Combining Deep Learning and Radiomics for Automated, Objective, Comprehensive Bone Marrow Characterization From Whole-Body MRI: A Multicentric Feasibility Study. Invest Radiol. 2022 Nov 1;57(11):752-763. doi: 10.1097/RLI.0000000000000891. Epub 2022 May 27. PMID 35640004
- [Derived] Wennmann M, Goldschmidt H, Mosebach J, Hielscher T, Bauerle T, Komljenovic D, McCarthy PL, Merz M, Schlemmer HP, Raab MS, Sauer S, Delorme S, Hillengass J. Whole-body magnetic resonance imaging plus serological follow-up for early identification of progression in smouldering myeloma patients to prevent development of end-organ damage. Br J Haematol. 2022 Oct;199(1):65-75. doi: 10.1111/bjh.18232. Epub 2022 May 24. PMID 35608264